CLINICAL TRIAL: NCT04562610
Title: A Prospective Study of Enhanced Recovery After Surgery in Orthopaedic Spine Surgery: Administration of Preoperative Oral Versus Intravenous Medications
Brief Title: Enhanced Recovery After Surgery in Orthopaedic Spine Surgery
Acronym: ERAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1586560
Record Dates: First submitted 2020-06-19; First posted 2020-09-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Surgery
Keywords: lumbar decompression and fusions 1 to 3 levels; lumbar decompression and fusions

STUDY DESIGN:
Intervention Model Description: The investigators are comparing the efficacy of commonly administered pre-emptive analgesic medications administered in a randomized fashion in parallel. In one group all medications will be administered by mouth and in one group two of the medications will be administered via the intravenous route.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: All oral pre-operative analgesics (Active Comparator): Group A patients will be administered the following medications in the preoperative holding area:
  * Acetaminophen 1,000 mg by mouth prior to operation
  * Celecoxib 200mg by mouth prior to operation
  * Tranexamic acid 2 grams by mouth prior to operation
  * Gabapentin 600mg by mouth prior to operation
  Interventions: Drug: All oral administration group
- Group B: Intravenous agents (Active Comparator): Group B patients will receive:
  * Acetaminophen (Ofirmev) 1,000mg intravenous prior to operation
  * Celecoxib 200mg by mouth prior to operation
  * Tranexamic acid 2grams intravenous at start of operation
  * Gabapentin 600 mg by mouth prior to operation
  Interventions: Drug: Intravenous Infusion group

INTERVENTIONS:
Drug: Intravenous Infusion group — The intravenous infusion group will receive two medications via the intravenous infusion route. These medications are Ofirmev ( acetaminophen ) 1,000mg and tranexamic acid 2,000 mg , an antifibrinolytic drug. In addition to these drugs, study subjects will receive Celecoxib 200mg by mouth and Gabapentin 600 mg by mouth prior to operation.
  Arms: Group B: Intravenous agents
Drug: All oral administration group — Subjects in the oral administration group will receive the following pre-emptive analgesic drugs, acetaminophen 1,000mg, Celecoxib 200mg and gabapentin 600mg via the oral route prior to operation. In addition they will receive the antifibrinolytic drug, tranexamic acid 2,000mg via an oral route as well prior to operation.
  Arms: Group A: All oral pre-operative analgesics

SUMMARY:
This study aims to determine the impact and effect of enhanced recovery after surgery (ERAS) principles in the recovery and rehabilitation of patients following elective orthopaedic spine surgery with a specific emphasis on oral versus intravenous preoperative medication administration and the resultant cost differences.

DETAILED DESCRIPTION:
In orthopaedic surgery, ERAS programs have profoundly impacted outcomes in hip and knee replacement surgery.4 Large, prospective studies have demonstrated a reduction in mortality rate, median length of stay, and blood transfusion rates with no change in re-admission rates.5,6 However, there is a paucity of data evaluating the application of ERAS principles in other orthopaedic subspecialties, especially elective spine surgery. With over 35,000 cervical spine procedures performed in 2011, almost 200,000 elective lumbar fusion surgeries performed in 2015, and 83.7 million people estimated to be ≥ 65 years old in 2050, the demand for elective spine surgery is high and will continue to grow placing a significant economic burden on the health care system.This increasing demand in conjunction with prolonged hospital stays, extensive postoperative pain regimens, and the advent of minimally invasive procedures provides a compelling argument for the suitability of ERAS protocols in elective spine surgery.

While distinct components of the ERAS pathway have been investigated in spine surgery including preoperative education, multimodal pain management, surgical approach, nutrition, and physical therapy, few studies have investigated the collective application of these interventions. Furthermore, these studies have been retrospective in nature, limiting their generalizability.The goal of this study is to perform a prospective, randomized trial to evaluate the efficacy and cost-effectiveness of oral versus intravenous medications preoperatively. The investigators also plan to evaluate the effect of the implementation of the standard of care ERAS principles on the outcome of patients undergoing elective spine surgery.

ELIGIBILITY:
Inclusion Criteria:

· Surgery scheduled for lumbar decompression and fusions 1 to 3 levels

Exclusion Criteria:

* Cervical, thoracic, or lumbar trauma
* Oncologic procedures
* Patient's with comorbidities preventing early postoperative mobilization
* Patients with contraindications to tranexamic acid (TXA) administration including but not limited to patients with a history of thromboembolic or ischemic events (PE, DVT, CVA, MI). Additional contraindications are decided by treating orthopaedic surgeon

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Operative blood loss (ml) | From incision start to wound closed. 0-6 hours after operation start.
  Actual or estimated blood loss during operation. This is typically included in the surgeons operative note.
Postoperative pain scores (VAS) Visual analog scale. | The investigators will measure change between baseline/pre-surgical VAS score to immediate post surgical VAS, and at 4 hour intervals until hospital discharge. 0-48 hours
  Visual analog pain score from 1-10 points reported by patient with 10 severe pain and 0 being no pain. The investigators are comparing the efficacy of two different analgesia regimens, this is a critical primary outcome measure.
Immediate postoperative opiate analgesic requirement | From post anesthesia care unit admission until hospital discharge. As the investigators are measuring the 24 hour Morphine equivalent dosing from anesthesia emergence until hospital discharge. ( 0-48 hours after operation)
  Immediate post procedure Opiate analgesic requirement measured in Morphine equivalents (mg)
Time from post-anesthesia care unit (PACU) admission to discharge | PACU admission to PACU discharge (range 0-6 hours)
  This is the time from anesthesia emergence to initiation of meaningful activity. and recovery measured from anesthetic (in hours) with a range of 1-12 hours.
blood transfusion requirement | At any time point during hospitalization. ( 0-48 hours after operation)
  Amount of blood transfused expressed in milliliters (ml). As this may range from binary ( yes or no ) and could also be recorded in volume milliliters; the owill record and report both.
Length of hospital stay | From day of operation (day zero) through hospital discharge.Expected range 1-3 days)
  Length of hospital stay (LOS) in days with a range from 1-6 days.

SECONDARY OUTCOMES:
Overall cost of hospitalization. | Admission to outpatient surgery until discharge from the hospital, range expected 6-72 hours.
  Total cost of hospitalization including hospital stay, pharmacy charges, and other professional fees.
Post operative complications | From initiation of operation to hospital discharge (Day1-3)
  This outcome will be binary (yes/no). The investigators will record the occurrence of any operative or postoperative complications from hospital admission to hospital discharge. If no complications occur these will be recorded as zero; should complications occur during hospitalization, these complication will be recorded (readmission rate, infection, wound dehiscence, return to OR, deep vein thrombosis/pulmonary embolism (DVT/PE). Intra-operative complications, postoperative complications, including but not limited to respiratory events, GI complications including ileus, postoperative nausea and vomiting, ground level falls, orthostatic hypotensive events or any complication associated with early mobilization. The number of complications will be listed in addition to the individual complication type.
Oswestry Disability Index (ODI) | The investigators will measure change between baseline (ODI) and at surgical visits and 12 months after operation.
  10 question survey instrument with domains which include pain, physical, and social function. The range of scores is from 0-100 with 0 being no disability and 100 representing bedbound patients with no capacity to function in any domain.
Patient Reported Outcome Measurement Information System, Computer Adaptive Tests (PROMIS CAT) | The investigators will measure change between PROMIS CAT scores between between baseline and 12 months after operation.
  NIH computer adapted technology patient reported outcomes measures of pain interference, physical function, depression, anxiety, and upper extremity function.
University of California, Davis Short Form 20 (UCD SF-20) | The investigators will measure change between baseline pre-op SF-20 scores and 12 months after operation
  Patient reported outcome instrument with 20 questions and score between range 0- 100 points. Domains surveyed include self perception of health, bodily pain, social function, physical function and role emotional health.

CONTACTS AND LOCATIONS:
Overall Officials: Rolando F Roberto, MD, Principal Investigator — Univeristy of California Davis Medical Center
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Carli F. Physiologic considerations of Enhanced Recovery After Surgery (ERAS) programs: implications of the stress response. Can J Anaesth. 2015 Feb;62(2):110-9. doi: 10.1007/s12630-014-0264-0. Epub 2014 Dec 12. PMID 25501695
- [Background] Wainwright TW, Immins T, Middleton RG. Enhanced recovery after surgery (ERAS) and its applicability for major spine surgery. Best Pract Res Clin Anaesthesiol. 2016 Mar;30(1):91-102. doi: 10.1016/j.bpa.2015.11.001. Epub 2015 Nov 23. PMID 27036606
- [Background] Starks I, Wainwright TW, Lewis J, Lloyd J, Middleton RG. Older patients have the most to gain from orthopaedic enhanced recovery programmes. Age Ageing. 2014 Sep;43(5):642-8. doi: 10.1093/ageing/afu014. Epub 2014 Mar 13. PMID 24627354
- [Background] Aasvang EK, Luna IE, Kehlet H. Challenges in postdischarge function and recovery: the case of fast-track hip and knee arthroplasty. Br J Anaesth. 2015 Dec;115(6):861-6. doi: 10.1093/bja/aev257. Epub 2015 Jul 25. PMID 26209853
- [Background] Marquez-Lara A, Nandyala SV, Fineberg SJ, Singh K. Current trends in demographics, practice, and in-hospital outcomes in cervical spine surgery: a national database analysis between 2002 and 2011. Spine (Phila Pa 1976). 2014 Mar 15;39(6):476-81. doi: 10.1097/BRS.0000000000000165. PMID 24365907
- [Background] Martin BI, Mirza SK, Spina N, Spiker WR, Lawrence B, Brodke DS. Trends in Lumbar Fusion Procedure Rates and Associated Hospital Costs for Degenerative Spinal Diseases in the United States, 2004 to 2015. Spine (Phila Pa 1976). 2019 Mar 1;44(5):369-376. doi: 10.1097/BRS.0000000000002822. PMID 30074971
- [Background] Ortman, Jennifer M, Velkoff, Victoria A, Hogan H. An Aging Nation: The Older Population in the United States. Washington DC; 2014.
- [Background] Smith J, Probst S, Calandra C, Davis R, Sugimoto K, Nie L, Gan TJ, Bennett-Guerrero E. Enhanced recovery after surgery (ERAS) program for lumbar spine fusion. Perioper Med (Lond). 2019 May 28;8:4. doi: 10.1186/s13741-019-0114-2. eCollection 2019. PMID 31149331
- [Background] Corniola MV, Debono B, Joswig H, Lemee JM, Tessitore E. Enhanced recovery after spine surgery: review of the literature. Neurosurg Focus. 2019 Apr 1;46(4):E2. doi: 10.3171/2019.1.FOCUS18657. PMID 31018257
- [Background] Angus M, Jackson K, Smurthwaite G, Carrasco R, Mohammad S, Verma R, Siddique I. The implementation of enhanced recovery after surgery (ERAS) in complex spinal surgery. J Spine Surg. 2019 Mar;5(1):116-123. doi: 10.21037/jss.2019.01.07. PMID 31032446
- [Background] Elsarrag M, Soldozy S, Patel P, Norat P, Sokolowski JD, Park MS, Tvrdik P, Kalani MYS. Enhanced recovery after spine surgery: a systematic review. Neurosurg Focus. 2019 Apr 1;46(4):E3. doi: 10.3171/2019.1.FOCUS18700. PMID 30933920
- [Background] de Castro SM, van den Esschert JW, van Heek NT, Dalhuisen S, Koelemay MJ, Busch OR, Gouma DJ. A systematic review of the efficacy of gum chewing for the amelioration of postoperative ileus. Dig Surg. 2008;25(1):39-45. doi: 10.1159/000117822. Epub 2008 Feb 21. PMID 18292660
- [Background] Ali ZS, Ma TS, Ozturk AK, Malhotra NR, Schuster JM, Marcotte PJ, Grady MS, Welch WC. Pre-optimization of spinal surgery patients: Development of a neurosurgical enhanced recovery after surgery (ERAS) protocol. Clin Neurol Neurosurg. 2018 Jan;164:142-153. doi: 10.1016/j.clineuro.2017.12.003. Epub 2017 Dec 8. PMID 29232645
- [Background] Bilku DK, Dennison AR, Hall TC, Metcalfe MS, Garcea G. Role of preoperative carbohydrate loading: a systematic review. Ann R Coll Surg Engl. 2014 Jan;96(1):15-22. doi: 10.1308/003588414X13824511650614. PMID 24417824
- See also: Learn more or sign up for the study here! — https://studypages.com/s/enhanced-recovery-after-surgery-in-orthopaedic-spine-surgery-624518/